CLINICAL TRIAL: NCT01027572
Title: Efficacy of Thalamic Stimulation in the Treatment of Patients in Vegetative State and Minimally Conscious State From at Least Six Months. A Pilot Study
Brief Title: Thalamic Stimulation of Patients in Vegetative or Minimally Conscious State
Acronym: CATS\
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Roberto Imberti, Fondazione IRCCS Policlinico S. Matteo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RILM
Record Dates: First submitted 2009-12-01; First posted 2009-12-08 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Vegetative State; Minimally Conscious State
Keywords: Vegetative state; Minimally conscious state; Thalamic stimulation
MeSH Terms: conditions — Persistent Vegetative State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalamic stimulation (Experimental): Patients in Vegetative or Minimally Conscious State
  Interventions: Device: Implantable neurostimulation system (Medtronic)

INTERVENTIONS:
Device: Implantable neurostimulation system (Medtronic) — Thalamic stimulation will be performed using an implantable neurostimulation system

SUMMARY:
Rationale. The investigators hypothesize that bilateral electrical central thalamic stimulation of patients in Vegetative State and Minimally Conscious State from at least 6 months could improve the level of responsiveness.

Aims. Evaluate the efficacy of bilateral electrical central thalamic stimulation in patients in Vegetative State and Minimally Conscious State.

Study Design. Patients in Vegetative State and Minimally Conscious State from at least 6 months because of traumatic brain injury, hypoxic or ischemic brain injury will be evaluated to confirm the diagnosis according to the recent literature criteria. Then patients will be investigated by magnetic resonance (MRI), EEG and evoked potentials to evaluate eligibility. Patients included into the study will be implanted with electrodes, targeting the centromedian/parafascicularis nucleus complex of the thalamus bilaterally.

In the following months patients will be repeatedly evaluated using the CRS-R and Coma/Near Coma scales and the neurophysiologic parameters (EEG, evoked potentials) to assess the effects of thalamic stimulation. fMRI,DTI and MRS will be performed prior and after thalamic stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients stably in VS or MCS from at least 6 months, 10 to 65 years old.
* Patients must fulfil the neuroimaging criteria described later
* Patients must fulfil neurophysiologic criteria as described later

Exclusion Criteria:

* Inability to provide the informed consent by the legal representative
* Age < 10 years and > 65 years
* Pregnancy
* Expected life span < 1 year
* Presence of infectious disease not treatable
* Brain pathology not correlated with VS or MCS

Inclusion criteria based on MRI imaging of the brain. The following criteria specify the location and extent of damage to the brain which determine the inclusion or exclusion from the study.

Before inclusion into the study all patients will be submitted to a complete MRI of the brain comprehensive of T1 and T2 weighted and flair sequences. Patients with a history of traumatic injury that were not submitted to cervical MRI at the time or after the initial injury will be submitted to a cervical MRI before admission to the study. A MRI scanner with field strength of at least 1.5 tesla will be used for imaging the brain and the cervical spinal cord. The volumetric extent of the damage will be estimated by using an image analysis program (e.g. IMAGE, NIH) after the neuroradiologist has traced the contour of the injured structures in all MRI images of the brain.

Thalamus: bilateral absence of damage of the centromedian/parafascicularis complex and of the entire area of the intralaminar nuclei. The remaining structures of the thalami should not be damaged for an extent greater than 40% of the total volume of the two thalami.

Frontal lobes: at least one lobe should not be damaged to an extent superior to 20% of the volume. Absence of lesion of the Broca's area in the left (or dominant) hemisphere.

Temporal lobes: absence of damage to the posterior two third of the left or dominant temporal lobe. The extent of the lesions in the remaining structures of the temporal lobes should be less than 70% of the total volume of the lobes.

Parietal lobes: lesion volume in at least one parietal lobe should be less than 30%.

Occipital lobes: lesion volume in at least one occipital lobe should be less than 30%. The visual cortex should be spared in at least one lobe.

Hypothalamus: absence of lesions. Mesencephalon: absence of lesions in the region located between the substantia nigra and the bases of the colliculi. Unilateral lesions ventral to the substantia nigra are permitted.

Pons: absence of lesions unless unilateral and limited to the ventral third of the pons.

Cerebellum: Absence of lesions larger than 80% of the total volume; the deep nuclei of at least one side of the cerebellum should be intact.

Medulla: absence of lesions unless limited to one pyramid. Cervical spinal cord: absence of lesions All patients should be free from hydrocephalus or the hydrocephalus should be treated with a shunt prior to thalamic implant.

Exclusion criteria based on MRI imaging of the brain. All patients who do not fulfill the criteria for inclusion based on MRI imaging of the brain will be excluded.

Inclusion Criteria based on neurophysiologic parameters

* Patients will be studied by continuous electroencephalography. Patients showing EEG desynchronization for at least 5% of the period studied will be included.
* Acoustic evoked potentials must be present at least at one side. V wave prolongation will be accepted.
* Somato-sensory evoked potentials must be present at least at one side. Increased latency of N20 will be accepted.

Exclusion Criteria based on neurophysiologic criteria All patients who do not fulfill the criteria for inclusion based on neurophysiologic parameters will be excluded.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of thalamic stimulation evaluated by the administration of the CRS-R and Coma/Near Coma scales and comparing the results obtained with those of the pre-implant evaluation. | 1, 6, 12 months

SECONDARY OUTCOMES:
Changes in the length of desynchronization performed by continuous EEG recording and spectral analysis. Evaluate which patients in Vegetative State and Minimally Conscious State can benefit from central thalamic stimulation. | 1, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Imberti, MD, Study Chair — Fondazione IRCCS Policlinico S. Matteo - Pavia - Italy; Lorenzo Magrassi, MD, Study Chair — Fondazione IRCCS Policlinico S. Matteo, Pavia and University of Pavia - Italy
Locations (3):
- Italy (3):
  - Istituto di Bioimmagini e Fisiologia Molecolare - CNR, Milan
  - Fondazione IRCCS "Casimiro Mondino", Pavia
  - Fondazione IRCCS "Salvatore Maugeri", Pavia

REFERENCES:
- [Background] Schiff ND, Giacino JT, Kalmar K, Victor JD, Baker K, Gerber M, Fritz B, Eisenberg B, Biondi T, O'Connor J, Kobylarz EJ, Farris S, Machado A, McCagg C, Plum F, Fins JJ, Rezai AR. Behavioural improvements with thalamic stimulation after severe traumatic brain injury. Nature. 2007 Aug 2;448(7153):600-3. doi: 10.1038/nature06041. PMID 17671503
- [Background] Lombardi F, Gatta G, Sacco S, Muratori A, Carolei A. The Italian version of the Coma Recovery Scale-Revised (CRS-R). Funct Neurol. 2007 Jan-Apr;22(1):47-61. PMID 17509244
- [Background] Yamamoto T, Kobayashi K, Kasai M, Oshima H, Fukaya C, Katayama Y. DBS therapy for the vegetative state and minimally conscious state. Acta Neurochir Suppl. 2005;93:101-4. doi: 10.1007/3-211-27577-0_17. PMID 15986737
- [Derived] Magrassi L, Maggioni G, Pistarini C, Di Perri C, Bastianello S, Zippo AG, Iotti GA, Biella GE, Imberti R. Results of a prospective study (CATS) on the effects of thalamic stimulation in minimally conscious and vegetative state patients. J Neurosurg. 2016 Oct;125(4):972-981. doi: 10.3171/2015.7.JNS15700. Epub 2016 Jan 8. PMID 26745476